CLINICAL TRIAL: NCT06739304
Title: The Effectiveness of Mindfulness-based Relapse Prevention: A Randomized Controlled Trial Study
Brief Title: The Effectiveness of Mindfulness-based Relapse Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U22A20302
Record Dates: First submitted 2023-11-30; First posted 2024-12-18 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-12

CONDITIONS: Substance Use Disorder
Keywords: addiction; Mindfulness-based Relapse Prevention; anxiety; depression; subliminal perception
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Relapse Prevention (Experimental): 250 adult USD females of Intervention group received the 8-week Group mindfulness intervention performed by psychiatrists，and were assessed three times, before, during(1-2 weeks after the MBI began), and after the intervention by a variety of clinical variables, cognitive task(reginal segmental task),fMRI and blood test to verify the effectiveness of the intervention method, attempting to expand the model of addiction and mindfulness.
  Interventions: Behavioral: Mindfulness-based Relapse Prevention
- Control group (No Intervention): the matched 250 females in Control group were assessed by the by a variety of clinical variables, cognitive task(reginal segmental task),FMRI and blood test.

INTERVENTIONS:
Behavioral: Mindfulness-based Relapse Prevention — 250 adult USD females of Intervention group received the 8-week Group mindfulness intervention performed by psychiatrists.
  Arms: Mindfulness-Based Relapse Prevention

SUMMARY:
This study developed a Mindfulness-based Relapse Prevention targeting craving. Based on the Randomized Controlled Trial design, 600 adult USD females and 600 adult USD males with methamphetamine, heroin, or ketamine in Intervention group(MBI) , the matched 250 subjects in Control group and 250 healthy matched controls (HC) participated in this study, 1200 adult USD subjects of Intervention group received the 8-week Group mindfulness intervention performed by psychiatrists. SUD patients were assessed three times, before, during(1-2 weeks after the MBI began), and after the intervention by a variety of clinical variables, cognitive task(reginal segmental task),fMRI and blood test to verify the effectiveness of the intervention method, attempting to expand the model of addiction and mindfulness.

DETAILED DESCRIPTION:
The Group Mindfulness-based intervention adhered to structured formal procedures, conducted by psychiatrists, and was scheduled once a week, where each session spans for two hours, interspersed with a 10-minute break. Starting from the second intervention, the previous intervention's contents and home practice were reviewed at the beginning of each subsequent intervention.

Based on the Randomized Controlled Trial design, the evaluation time nodes for clinical variables, cognitive task(reginal segmental task),fMRI and blood test were baseline (before intervention), 1-2 weeks after intervention began, and after intervention. All clinical variable scales were presented in paper form, the questions were clearly explained by researchers.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for DSM-5 of substance use disorders;
2. The duration of using the addictive substance shall not be less than 1 year;
3. Prohibit addictive substances for at least 48 hours before conducting magnetic resonance imaging scans;
4. Han nationality, junior high school or above education level, aged 18-57 years old;
5. Informed and agreed to participate in this study, with the consent of the Ethics Committee.

Exclusion Criteria:

1. Have a history of mental illness before taking drugs;
2. Other substance use disorders (excluding nicotine);
3. Brain organic diseases, history of craniocerebral injury, history of coma;
4. Individuals with mental disorders who meet the DSM-5 diagnostic criteria within two generations;
5. History of endocrine diseases; Those with abnormal function in blood, heart, liver, and kidney after examination;
6. Intelligence impairment IQ.

Ages: 25 Years to 57 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 1200 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-08-05 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-Depression Scale (PHQ-9) | before, during(1-2 weeks after the mindfulness-based intervention began), and immediately after the intervention
  A quick depression assessment. The minimum score is 0 and maximum is 27. Higher scores indicate higher levels of depression. Minimal depression: scores 1-4. Mild depression: scores 5-9. Moderate depression: scores 10-14. Moderately severe depression: 15-19. Severe depression: 20-27.
Beck Anxiety Inventory (BAI-21) | before, during(1-2 weeks after the mindfulness-based intervention began), and immediately after the intervention
  Anxiety Assessment with 21 items. Minimum score is 0, and maximum is 63. The higher scores indicate higher levels of anxiety.
region segmental task | before and immediately after the mindfulness-based intervention
  correct rate of reginal segmental task
fMRI | before, during(1-2 weeks after the mindfulness-based intervention began), and immediately after the intervention
  Brain structure and brain function

CONTACTS AND LOCATIONS:
Overall Officials: Yanhui Liao, MD, Study Director — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Due to ethical and privacy consideration, IPD might not be shared

REFERENCES:
- [Result] Carroll KM, Kiluk BD. Cognitive behavioral interventions for alcohol and drug use disorders: Through the stage model and back again. Psychol Addict Behav. 2017 Dec;31(8):847-861. doi: 10.1037/adb0000311. Epub 2017 Aug 31. PMID 28857574
- [Result] Da Silva Roggi P M, Da Gama M F N, Neves F S, et al. Update on treatment of craving in patients with addiction using cognitive behavioral therapy
- [Result] Mohan UR, Watrous AJ, Miller JF, Lega BC, Sperling MR, Worrell GA, Gross RE, Zaghloul KA, Jobst BC, Davis KA, Sheth SA, Stein JM, Das SR, Gorniak R, Wanda PA, Rizzuto DS, Kahana MJ, Jacobs J. The effects of direct brain stimulation in humans depend on frequency, amplitude, and white-matter proximity. Brain Stimul. 2020 Sep-Oct;13(5):1183-1195. doi: 10.1016/j.brs.2020.05.009. Epub 2020 May 21. PMID 32446925
- [Result] Solinas M, Belujon P, Fernagut PO, Jaber M, Thiriet N. Dopamine and addiction: what have we learned from 40 years of research. J Neural Transm (Vienna). 2019 Apr;126(4):481-516. doi: 10.1007/s00702-018-1957-2. Epub 2018 Dec 19. PMID 30569209
- [Result] Hare BD, Duman RS. Prefrontal cortex circuits in depression and anxiety: contribution of discrete neuronal populations and target regions. Mol Psychiatry. 2020 Nov;25(11):2742-2758. doi: 10.1038/s41380-020-0685-9. Epub 2020 Feb 21. PMID 32086434
- [Result] Wydra K, Suder A, Frankowska M, Borroto Escuela DO, Fuxe K, Filip M. Effects of intra-accumbal or intra-prefrontal cortex microinjections of adenosine 2A receptor ligands on responses to cocaine reward and seeking in rats. Psychopharmacology (Berl). 2018 Dec;235(12):3509-3523. doi: 10.1007/s00213-018-5072-8. Epub 2018 Nov 13. PMID 30426181
- [Result] Feil J, Zangen A. Brain stimulation in the study and treatment of addiction. Neurosci Biobehav Rev. 2010 Mar;34(4):559-74. doi: 10.1016/j.neubiorev.2009.11.006. Epub 2009 Nov 13. PMID 19914283
- [Result] Hoppes K. The application of mindfulness-based cognitive interventions in the treatment of co-occurring addictive and mood disorders. CNS Spectr. 2006 Nov;11(11):829-51. doi: 10.1017/s1092852900014991. PMID 17075556
- [Result] Chen P, Jindani F, Perry J, et al. Mindfulness and problem gambling treatment
- [Result] Grant S, Colaiaco B, Motala A, Shanman R, Booth M, Sorbero M, Hempel S. Mindfulness-based Relapse Prevention for Substance Use Disorders: A Systematic Review and Meta-analysis. J Addict Med. 2017 Sep/Oct;11(5):386-396. doi: 10.1097/ADM.0000000000000338. PMID 28727663
- [Result] Witkiewitz K, Lustyk MKB, Bowen S. Retraining the addicted brain: a review of hypothesized neurobiological mechanisms of mindfulness-based relapse prevention. Psychol Addict Behav. 2013 Jun;27(2):351-365. doi: 10.1037/a0029258. Epub 2012 Jul 9. PMID 22775773
- [Result] Chambers R, Lo B C Y, Allen N B. The impact of intensive mindfulness training on attentional control, cognitive style, and affect
- [Result] Bowen S, Chawla N, Collins SE, Witkiewitz K, Hsu S, Grow J, Clifasefi S, Garner M, Douglass A, Larimer ME, Marlatt A. Mindfulness-based relapse prevention for substance use disorders: a pilot efficacy trial. Subst Abus. 2009 Oct-Dec;30(4):295-305. doi: 10.1080/08897070903250084. PMID 19904665
- [Result] Winhall J. Treating trauma and addiction with the felt sense polyvagal model: A bottom-up approach
- [Result] Froeliger B, McConnell PA, Stankeviciute N, McClure EA, Kalivas PW, Gray KM. The effects of N-Acetylcysteine on frontostriatal resting-state functional connectivity, withdrawal symptoms and smoking abstinence: A double-blind, placebo-controlled fMRI pilot study. Drug Alcohol Depend. 2015 Nov 1;156:234-242. doi: 10.1016/j.drugalcdep.2015.09.021. Epub 2015 Sep 26. PMID 26454838
- [Result] Garland EL. Restructuring reward processing with Mindfulness-Oriented Recovery Enhancement: novel therapeutic mechanisms to remediate hedonic dysregulation in addiction, stress, and pain. Ann N Y Acad Sci. 2016 Jun;1373(1):25-37. doi: 10.1111/nyas.13034. Epub 2016 Apr 1. PMID 27037786
- [Result] Garland E L, Bryan M A, Hanley A W, et al. Neurocognitive mechanisms of mindfulness-based interventions for addiction
- [Result] Garland EL, Froeliger B, Howard MO. Effects of Mindfulness-Oriented Recovery Enhancement on reward responsiveness and opioid cue-reactivity. Psychopharmacology (Berl). 2014 Aug;231(16):3229-38. doi: 10.1007/s00213-014-3504-7. Epub 2014 Mar 5. PMID 24595503
- [Result] Kirlic N, Cohen Z, Stewart J L. Neurocircuitry of Mindfulness-Based Interventions for Substance Use Prevention and Recovery
- [Result] Parks G A, Marlatt G A. Relapse prevention therapy: A cognitive-behavioral approach
- [Result] Witkiewitz K, Marlatt G A, Walker D. Mindfulness-based relapse prevention for alcohol and substance use disorders
- [Result] Ramos LA, Blankers M, van Wingen G, de Bruijn T, Pauws SC, Goudriaan AE. Predicting Success of a Digital Self-Help Intervention for Alcohol and Substance Use With Machine Learning. Front Psychol. 2021 Sep 3;12:734633. doi: 10.3389/fpsyg.2021.734633. eCollection 2021. PMID 34552539
- [Result] Knudsen HK, Abraham AJ, Roman PM. Adoption and implementation of medications in addiction treatment programs. J Addict Med. 2011 Mar;5(1):21-7. doi: 10.1097/ADM.0b013e3181d41ddb. PMID 21359109
- [Result] Sofuoglu M, DeVito EE, Waters AJ, Carroll KM. Cognitive Function as a Transdiagnostic Treatment Target in Stimulant Use Disorders. J Dual Diagn. 2016;12(1):90-106. doi: 10.1080/15504263.2016.1146383. PMID 26828702
- [Result] Friedman NP, Robbins TW. The role of prefrontal cortex in cognitive control and executive function. Neuropsychopharmacology. 2022 Jan;47(1):72-89. doi: 10.1038/s41386-021-01132-0. Epub 2021 Aug 18. PMID 34408280
- [Result] Lindgren KP, Hendershot CS, Ramirez JJ, Bernat E, Rangel-Gomez M, Peterson KP, Murphy JG. A dual process perspective on advances in cognitive science and alcohol use disorder. Clin Psychol Rev. 2019 Apr;69:83-96. doi: 10.1016/j.cpr.2018.04.002. Epub 2018 Apr 11. PMID 29680185
- [Result] Bradizza CM, Stasiewicz PR, Paas ND. Relapse to alcohol and drug use among individuals diagnosed with co-occurring mental health and substance use disorders: a review. Clin Psychol Rev. 2006 Mar;26(2):162-78. doi: 10.1016/j.cpr.2005.11.005. Epub 2006 Jan 6. PMID 16406196
- [Result] Perales JC, King DL, Navas JF, Schimmenti A, Sescousse G, Starcevic V, van Holst RJ, Billieux J. Learning to lose control: A process-based account of behavioral addiction. Neurosci Biobehav Rev. 2020 Jan;108:771-780. doi: 10.1016/j.neubiorev.2019.12.025. Epub 2019 Dec 14. PMID 31846653
- [Result] Diana M, Raij T, Melis M, Nummenmaa A, Leggio L, Bonci A. Rehabilitating the addicted brain with transcranial magnetic stimulation. Nat Rev Neurosci. 2017 Nov;18(11):685-693. doi: 10.1038/nrn.2017.113. Epub 2017 Sep 29. PMID 28951609
- [Result] Taylor AMW. Corticolimbic circuitry in the modulation of chronic pain and substance abuse. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Dec 20;87(Pt B):263-268. doi: 10.1016/j.pnpbp.2017.05.009. Epub 2017 May 10. PMID 28501595